CLINICAL TRIAL: NCT01573429
Title: Bisphenol A (BPA) Pharmacokinetic (PK): Controlled Exposure Study
Brief Title: Bisphenol A Controlled Exposure Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 120089; 12-E-0089
Record Dates: First submitted 2012-04-04; First posted 2012-04-09 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: Biologic Sample Collection; Metabolism; Healthy Volunteer; HV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dermal Carboxymethylcellulose arm (Other): d-BPA administered dermally using a carboxymethylcellulose suspension
  Interventions: Other: deuterated-Bisphenol A (d-BPA)
- Dermal ethanol arm (Other): d-BPA is administered dermally using an ethanol solution
  Interventions: Other: deuterated-Bisphenol A (d-BPA)
- Oral arm (Other): d-BPA administered orally
  Interventions: Other: deuterated-Bisphenol A (d-BPA)

INTERVENTIONS:
Other: deuterated-Bisphenol A (d-BPA) — The primary endpoints are key pharmacokinetic measurements of d-BPA and d-BPA conjugates in blood and urine over 6 days after a single dose of oral and/or ethanol solution dermal application and/or a carboxymethylcellulose suspension dermal application of a dose of 100 micro g/kg bw of d-BPA.

SUMMARY:
Background:

- Bisphenol A (BPA) is a chemical that is used primarily to make plastics, resins, and thermal paper. Most people are exposed daily to low levels of BPA that leaches into food and water from plastic products, including water and baby bottles. However, not all of the risks of BPA are known. Researchers want to learn more about how BPA acts in the body, and how the body gets rid of BPA.

Objectives:

- To study controlled exposure to BPA and its effects on the body.

Eligibility:

- Healthy, non-obese volunteers between 25 and 45 years of age.

Design:

* Participants will have six visits over about 2 to 4 weeks for this study.
* At the first visit, participants will be screened with a physical exam and blood and urine tests. They will complete a questionnaire about exposure to BPA-containing products. They will also receive a list of medications that should not be taken during the study period.
* The second visit will last about 13 hours. Participants will fast for 8 hours before the visit. They will then have a single dose of d-BPA (a modified form of BPA that is easier to study in the body). Regular blood samples will be taken over the 13-hour visit. All urine will also be collected. Participants will receive breakfast and lunch during the visit.
* Participants will have four follow-up visits. They will collect and store all of their urine between each follow-up visit. Blood samples will be collected at the follow-up visits....

DETAILED DESCRIPTION:
Bisphenol A (BPA) is utilized primarily in the manufacture of polycarbonate plastic and epoxy resins, which are widely used in the fabrication of baby bottles and food can linings. Consequently, human exposures to BPA are widespread. However, there is still uncertainty about the extent and nature of these exposures. This pharmacokinetic (PK) study is aimed at refining our understanding of the metabolism and excretion of BPA following two different routes of administration. This investigation is also intended to help resolve current controversies in BPA risk assessment. We will administer 100 microgram/kg body weight (bw) of deuterated BPA (d-BPA) orally and/or dermally (as an ethanol solution or a carboxymethylcellulose suspension), in up to 50 participants, with comparable numbers of men to women, and collect blood and urine for measurements of d-BPA and d-BPA conjugates at selected time points over a six day period post-dosing. The use of d-BPA will allow the detection of the administered BPA to be distinguished from background BPA. The primary endpoint of the study is detection of measurable d-BPA and d-BPA conjugates in blood and urine after administration of a single dose of 100 microgram/kg bw d-BPA applied orally and/or dermally (as an ethanol solution or a carboxymethylcellulose suspension). Participants will be given an option to complete either one or both phases of the study, the exposure visits separated by a period of at least 4 weeks. Dose selection was based on balancing the need for detectable levels of BPA in blood and urine to meet the objective and the need to minimize human subject risk. Data from the first 3 participants in the study, who received oral d-BPA, confirmed dosing during the oral pilot phase was sufficient in capturing measurable d-BPA in blood and urine and will continue at 100 microgram/kg bw of d-BPA for oral dosing. Dermal exposure will consist of a pilot phase for this route of administration comprising 4 participants to assess whether 100 microgram/kg bw of d-BPA applied to the skin is sufficient to obtain measurable d-BPA in blood and/or urine in order to establish PK parameters and to evaluate whether the time points are appropriate and necessary. If needed, the dermal pilot phase will be repeated using an ethanol solution rather than a carboxymethylcellulose suspension. The design includes sufficient sampling of blood and urine to define relevant PK parameters, including the rate of BPA absorption, plasma elimination rate, area under the curve (AUC) and apparent clearance, half-life, the urinary excretion rate, and the fractional metabolic clearance of the glucuronide and sulfate conjugates.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants meeting all of the following criteria will be considered for admission into this study:

* Male or female 25-45 years of age at the time of enrollment.
* Able to fast overnight (at least 8 hours).
* Able to understand and provide written informed consent in English.
* Able to travel to the NIEHS Clinical Research Unit (CRU) for all required study visits.
* Male and females of reproductive age agree to use contraception to avoid conceiving a child and agree not to donate eggs or sperm for six months following their participation in the study.

EXCLUSION CRITERIA:

* Uncontrolled diabetes:

  --Hemoglobin A1C of greater than or equal to 6.5% or a fasting blood glucose of greater than or equal to 126 mg/dL.
* Known liver dysfunction or disease:

  * ALT - higher than the normative value or determined abnormal by the PI.
  * AST - higher than the normative value or determined abnormal by the PI.
  * ALP - higher than the normative value or determined abnormal by the PI.
* Known kidney dysfunction or disease:

  * Estimated Glomerular Filtration Rate (eGFR)- <60 ml/min per the MDRD equation.
  * Clinically relevant anemia as defined as hemoglobin concentration <13g/dL for males and hemoglobin concentration <11g/dL for females.
* Pregnancy: Positive serum quantitative hCG pregnancy test.
* Current lactation.
* BMI less than or equal to 19 and greater than or equal to 35
* Medication use: Given the widespread use of medications, it may not be practical to instruct subjects to avoid all medication prior to and during the study. Thus, participant exclusion will be based on use of medications within 48 hours of the exposure and for the 6 days following the exposure that affect glucuronidation of the d-BPA dosage: Salicylic acid, acetaminophen, ibuprofen, naproxen, mefenamic acid, diclofenac, gliclazide carbamazepine, valproic acid, cimetidine, sulfasalazine, amoxicillin and erythromycin.
* Recent blood donation within the past 8 weeks of the BPA exposure visit (so as not to exceed donation of 10.5 mL/kg or 550 mL over an 8 week period).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07-18 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of d-BPA and d-BPA conjugates in blood and urine over 6 days | 6 days
  The primary endpoints are key pharmacokinetic measurements of d-BPA and d-BPA conjugates in blood and urine over 6 days after a single dose of oral and/or ethanol solution dermal application and/or acarboxymethylcellulose suspension dermal application of a dose of 100 micro g/kg bw of d-BPA.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Garantziotis, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-E-0089.html